CLINICAL TRIAL: NCT07010393
Title: A Multicenter Prospective-Retrospective Real-World Study Evaluating Conversion-to-Surgery and Survival After Genotype-Matched Neoadjuvant Systemic Therapy in Locally Advanced Thyroid Carcinoma
Brief Title: Genotype-Driven Neoadjuvant Therapy for Locally Advanced Thyroid Cancer: A Real-World Cohort Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Real-Neo
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Neoplasms
Keywords: Locally Advanced; Neoadjuvant Therapy; Real-World Study; BRAF V600E; RET Fusion; VEGF-TKI; Immunotherapy; Conversion Surgery; R0 Resection; Precision Oncology; Real-World Evidence; Conversion Therapy
MeSH Terms: conditions — Thyroid Neoplasms | interventions — dabrafenib; trametinib; selpercatinib; pralsetinib; lenvatinib; larotrectinib; anlotinib; pembrolizumab; sintilimab; cabozantinib; Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: Participants are assigned to seven genotype- or immunophenotype-defined, parallel, non-overlapping arms with no planned cross-over:
  Arm 1 (BRAF V600E) - dabrafenib + trametinib
  Arm 2 (RET fusion) - selpercatinib
  Arm 3 (RET point-mutation MTC) - selpercatinib or retrospective cohort on pralsetinib
  Arm 4 (NTRK fusion) - larotrectinib
  Arm 5 (TERT-only, driver-negative for BRAF/RET) - lenvatinib, anlotinib, or cabozantinib
  Arm 6 (Triple-negative, no actionable driver) - investigator-choice MKI (lenvatinib, anlotinib, cabozantinib)
  Arm 7 (PD-L1 ≥ 1 % or MKI-refractory) - PD-1/PD-L1 blockade (pembrolizumab, sintilimab, or domestic PD-L1 antibody bemosuzumab) ± MKI combination (e.g., pembrolizumab + lenvatinib) per treating physician
  Assignment is open-label, non-randomized; placement into an arm is decided before first dose by a central molecular & PD-L1 board reviewing NGS/PCR and IHC results. No cross-over permitted.
Masking Description: Assignment is open-label, non-randomized; placement into an arm is decided before first dose by a central molecular & PD-L1 board reviewing NGS/PCR and IHC results. No cross-over permitted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- BRAF V600E Mutation (Experimental): Dabrafenib 150 mg PO BID + trametinib 2 mg PO QD given in 28-day cycles (Day 1-28). After Cycle 4 (Day 112 ± 7) patients undergo imaging review; if previously unresectable disease becomes operable, conversion surgery is scheduled within 3 weeks. Those still unresectable continue treatment until progression/toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Lenvatinib; Drug: Anlotinib; Drug: Cabozantinib; Procedure: Conversion Surgery
- RET Fusion PTC (Experimental): Selpercatinib 160 mg PO BID, continuous 28-day cycles. Surgery conversion assessment at Day 112 (end of Cycle 4). Resectable cases proceed to thyroidectomy ± neck dissection; others maintain therapy per label.
  Interventions: Drug: Selpercatinib; Drug: Pralsetinib; Drug: Lenvatinib; Drug: Anlotinib; Drug: Cabozantinib; Procedure: Conversion Surgery
- RET Point-Mutation MTC (Experimental): Prospective cohort: selpercatinib 160 mg PO BID, 28-day cycles; Retrospective sub-cohort: historical pralsetinib 400 mg PO QD (also 28-day cycles). Cycle 4 reassessment (Day 112) for potential curative resection of residual neck disease or distant oligometastases.
  Interventions: Drug: Selpercatinib; Drug: Lenvatinib; Drug: Anlotinib; Drug: Cabozantinib; Procedure: Conversion Surgery
- NTRK Fusion (Experimental): Larotrectinib 100 mg PO BID in continuous 28-day cycles with multidisciplinary resectability evaluation after 4 cycles (Day 112). Eligible patients undergo surgery; non-eligible continue TRK inhibitor.
  Interventions: Drug: Lenvatinib; Drug: Larotrectinib; Drug: Anlotinib; Drug: Cabozantinib; Procedure: Conversion Surgery
- TERT-Only (MKI) (Experimental): Investigator-selected MKI: lenvatinib 24 mg PO QD (28-day cycle), anlotinib 12 mg PO d1-14 q21d (21-day cycle; Cycle 4 ends Day 84), or cabozantinib 60 mg PO QD (28-day cycle). Conversion-surgery review: Day 112 for 28-day regimens or Day 84 for anlotinib.
  Interventions: Drug: Lenvatinib; Drug: Anlotinib; Drug: Pembrolizumab; Drug: Sintilimab; Drug: Cabozantinib; Drug: Bemosuzumab; Procedure: Conversion Surgery
- Triple-Negative (driver-negative) - MKI (Experimental): Same MKI options/cycle lengths as Arm 5. Cycle 4 resectability check (Day 112 or Day 84 depending on drug). Successful conversions proceed to definitive surgery; others remain on systemic therapy.
  Interventions: Drug: Trametinib; Drug: Lenvatinib; Drug: Anlotinib; Drug: Pembrolizumab; Drug: Sintilimab; Drug: Cabozantinib; Drug: Bemosuzumab; Procedure: Conversion Surgery
- PD-L1 ≥ 1 % / MKI-Refractory - Immunotherapy ± MKI (Experimental): Checkpoint agents: pembrolizumab 200 mg IV q3w (21-day cycles), sintilimab 200 mg IV q3w (21 d), or domestic PD-L1 Ab bemosuzumab 900 mg IV q2w (14-day cycles). Combination option: lenvatinib 20 mg PO QD (28-day cycles) added at investigator discretion. Conversion assessment occurs after 4 cycles of the longest component being used (e.g., Day 84 for pembrolizumab; Day 112 if combined with 28-day MKI). Resectable patients undergo surgery; others continue or switch therapy.
  Interventions: Drug: Lenvatinib; Drug: Anlotinib; Drug: Pembrolizumab; Drug: Sintilimab; Drug: Cabozantinib; Drug: Bemosuzumab; Procedure: Conversion Surgery

INTERVENTIONS:
Drug: Dabrafenib — 150 mg orally twice daily; ≤4 × 28-day cycles
  Arms: BRAF V600E Mutation
Drug: Trametinib — 2 mg orally once daily; same duration
  Arms: BRAF V600E Mutation; Triple-Negative (driver-negative) - MKI
Drug: Selpercatinib — 160 mg orally twice daily; ≤4 cycles
  Arms: RET Fusion PTC; RET Point-Mutation MTC
Drug: Pralsetinib — retrospective, 400 mg orally once daily; ≤4 cycles
  Arms: RET Fusion PTC
Drug: Lenvatinib — 24 mg orally once daily; ≤4 cycles
Drug: Larotrectinib — Larotrectinib 100 mg orally twice daily, continuous 28-day cycles.
  Arms: NTRK Fusion
Drug: Anlotinib — 12 mg orally once daily; 2 weeks on / 1 week off, ≤4 cycles (alternative)
Drug: Pembrolizumab — 200 mg IV infusion every 3 weeks; ≤4 cycles
  Arms: PD-L1 ≥ 1 % / MKI-Refractory - Immunotherapy ± MKI; TERT-Only (MKI); Triple-Negative (driver-negative) - MKI
Drug: Sintilimab — 200 mg IV infusion every 3 weeks; ≤4 cycles
  Arms: PD-L1 ≥ 1 % / MKI-Refractory - Immunotherapy ± MKI; TERT-Only (MKI); Triple-Negative (driver-negative) - MKI
Drug: Cabozantinib — Cabozantinib 60 mg orally once daily, continuous 28-day cycles.
Drug: Bemosuzumab — China PD-L1 antibody bemosuzumab 900 mg IV every 2 weeks (14-day cycle).
  Arms: PD-L1 ≥ 1 % / MKI-Refractory - Immunotherapy ± MKI; TERT-Only (MKI); Triple-Negative (driver-negative) - MKI
Procedure: Conversion Surgery — Conversion Surgery if resectable

SUMMARY:
This multicenter registry tests whether genomically matched neoadjuvant therapy (1-4 cycles tailored to BRAF V600E, RET fusion/mutation, isolated TERT mutation, triple-negative BRAF/RET/TERT, or ICI ± TKI) can render locally advanced, initially unresectable-or high-morbidity-thyroid cancers operable. The primary endpoint is conversion-to-surgery; key secondaries are R0/1 margin rate and 12-month event-free survival, with propensity-score weighting correcting cohort imbalances. Findings aim to define a precision-guided neoadjuvant standard for down-staging advanced thyroid tumors.

DETAILED DESCRIPTION:
This multicenter, prospective-retrospective registry will determine whether genotype-matched neoadjuvant systemic therapy can convert locally advanced, initially unresectable or high-morbidity thyroid cancers to successful surgery. Patients receive one to four 28-day cycles of treatment chosen according to actionable genomic alterations-BRAF V600E, RET fusion, RET point mutation, isolated TERT promoter mutation, "BRT triple-negative" (wild-type for BRAF/RET/TERT), or immune-checkpoint blockade ± TKI-before reassessment by a multidisciplinary team.

Primary outcome is the conversion-to-surgery rate. Key secondary outcomes include R0/1 (margin-negative) resection rate and 12-month event-free survival, defined as absence of progression, unresectability at planned surgery, recurrence, or death. Propensity-score weighting will balance baseline differences among cohorts and permit adjusted comparisons. Results will clarify the role of targeted and immunologic agents in down-staging advanced thyroid tumors and may establish a precision-guided neoadjuvant standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at enrollment.
2. Histologically or cytologically confirmed thyroid carcinoma that meets ≥ 1 of the following:

   * Radioactive-iodine-refractory differentiated thyroid carcinoma (DTC)
   * Medullary thyroid carcinoma (MTC)
   * Anaplastic or poorly differentiated thyroid carcinoma (ATC/PDTC)
   * Other locally advanced / metastatic thyroid malignancy deemed incurable by surgery alone.
3. Disease judged unresectable or entailing prohibitively high-morbidity surgery at baseline by a multidisciplinary thyroid-oncology board.
4. Documented molecular or immunophenotype qualifying for ≥ 1 study arm:

   * BRAF V600E mutation
   * RET gene fusion
   * RET activating point mutation (e.g., M918T)
   * NTRK1/2/3 fusion
   * Isolated TERT-promoter mutation with no BRAF/RET/NTRK alterations
   * Driver-negative / VEGFR-wild type ("triple-negative")
   * PD-L1 expression ≥ 1 % OR progression after prior multi-kinase inhibitor (MKI).
5. ECOG Performance Status 0-2.
6. At least one measurable lesion per RECIST v1.1 / iRECIST (MTC with calcitonin/CEA evaluable disease accepted).
7. Written informed consent obtained.

Exclusion Criteria:

1. Untreated or symptomatic CNS metastases; patients with treated, stable lesions ≥ 4 weeks and off corticosteroids are eligible.
2. Pregnant or breastfeeding. Women and men of child-bearing potential must agree to effective contraception during study and for ≥ 120 days after last dose (≥ 180 days for men after dabrafenib/trametinib).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-World Progression-Free Survival (rwPFS) | Baseline to radiologic/clinical progression or death, whichever occurs first, up to 36 months
  Time from Cycle 1 Day 1 to the earliest date of disease progression (RECIST/iRECIST) or all-cause death.

SECONDARY OUTCOMES:
Real-World Objective Response Rate (rwORR) | Baseline to first documented response, assessed every 8-12 weeks, up to 24 months
  Percentage of patients with complete or partial response per RECIST v1.1 (or iRECIST for immunotherapy arms) as determined by local radiology.
Pathologic Tumor Regression ≥ 50 % | At surgery
  Proportion of surgical specimens showing ≥ 50 % reduction in viable tumor area compared with baseline imaging estimate.
R0/1 Resection Rate | At surgery (≈ 1-5 months after first dose)
  Percentage of resected participants whose final pathology shows microscopically negative (R0) or close (R1 ≤ 1 mm) margins.
Conversion-to-Surgery Rate | Up to 12 months from first dose
  Proportion of enrolled participants who proceed to the intended curative-intent resection after completion of neoadjuvant therapy.
Overall Survival (OS) | Baseline to death from any cause, censored at 36 months
  Time from Cycle 1 Day 1 to death; survivors censored at last known follow-up.
Duration of Response (DoR) | From first documented response until progression or death, up to 36 months
  Among responders, time between initial response and subsequent disease progression or death.
Incidence of Grade ≥ 3 Treatment-Related AEs | Baseline to 30 days after last dose
  Number and percentage of participants experiencing Grade 3 or higher adverse events per CTCAE v5.0.
Quality-of-Life Change (EORTC QLQ-THY34) | Baseline, pre-surgery, and 6 months post-surgery
  Mean change from baseline in global QoL score.
Thyroglobulin Reduction ≥ 90 % | Pre-surgery (≈ 4 months)
  Proportion of differentiated-tumor participants with ≥ 90 % decrease in serum thyroglobulin from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
De-identified datasets will be available 6 months after primary publication via institutional repository upon reasonable request